CLINICAL TRIAL: NCT00514384
Title: Prognostic Value of Serial Biomarker Measurements in Patients With ADHF
Brief Title: Serial Measurements of Biomarker in Patients With Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Serial Biomarker in ADHF
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of serial measurement of novel biomarker for diagnosis, prognosis or therapy monitoring in patients presenting with acute decompensated heart failure.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a chronic and progressive illness resulting from a variety of cardiac causes, including ischemic and valvular heart disease, dilatative cardiomyopathy or hypertension. HF may also develop suddenly, particularly as a complication of acute myocardial infarction or as an acute exacerbation in patients with previously compensated chronic HF. Diagnosis and in-hospital management of HF is often demanding and outcome especially regarding rehospitalizations is impaired. Novel biomarker may be very helpful in assessment of diagnosis, prognosis, and severity of HF as well as for treatment monitoring.

Design: Prospective, multicenter observational study Setting: University Hospital Basel, Kantonsspital Aarau, Kantonsspital Luzern, Kantonsspital Wolhusen Patients: Patients with acute HF not requiring ICU admission

Measurement of serial biomarker (BNP, NT-proBNP, MR-proADM, ST2, hs-cTnI and Copeptin) will be performed at presentation, at 6 hours (h), 12h, 18h, 24h, at 48h, at day 6 and at hospital discharge. Follow- up will be performed at 6 Month, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute HF
* Informed consent

Exclusion Criteria:

* Cardiogenic shock, ST-elevation myocardial infarction, or other clinical conditions that require immediate ICU admission or urgent PTCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ADHF not requiering ICU
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2007-02; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Course of BNP, NT-proBNP, MR-proADM, Copeptin, ST2, hsTnT | Entry, 6h, 12h, 18h, 24h, 48h, 6 days, discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mueller Christian, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (4):
- Switzerland (4):
  - Cantonal Hospital Aarau, Aarau, Canton of Aargau
  - University Hospital Lucerne, Lucerne, Canton of Lucerne
  - Hospital Wolhusen, Wolhusen, Canton of Lucerne
  - University Hospital Basel, Basel

REFERENCES:
- [Derived] Noveanu M, Breidthardt T, Potocki M, Reichlin T, Twerenbold R, Uthoff H, Socrates T, Arenja N, Reiter M, Meissner J, Heinisch C, Stalder S, Mueller C. Direct comparison of serial B-type natriuretic peptide and NT-proBNP levels for prediction of short- and long-term outcome in acute decompensated heart failure. Crit Care. 2011;15(1):R1. doi: 10.1186/cc9398. Epub 2011 Jan 5. PMID 21208408